CLINICAL TRIAL: NCT04213404
Title: Ribociclib and Spartalizumab for Head and Neck Squamous Cell Carcinoma, a Phase I Study With Expansion Cohort (RISE-HN)
Brief Title: Ribociclib and Spartalizumab in R/M HNSCC
Acronym: RISE-HN
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201907017MIPD; CPDR001A0TW01T (Other Grant/Funding Number: Novartis); RISE-HN (Other: Taiwan FDA)
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: ribociclib; spartalizumab; PDR001; head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — ribociclib; spartalizumab

STUDY DESIGN:
Intervention Model Description: single arm, phase I study with dose titration plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ribociclib-spartalizumab (Experimental): Ribociclib 400mg, 600mg, or 200mg oral daily, D1-D21, 28 days a cycle Spartalizumab 400mg ivdrip on D1, 28 days a cycle.
  Interventions: Drug: Ribociclib; Drug: Spartalizumab

INTERVENTIONS:
Drug: Ribociclib — Ribociclib 400mg, 600mg, or 200mg oral daily, D1-D21, 28 days a cycle
  Other Names: Kisqali
Drug: Spartalizumab — Spartalizumab 400mg ivdrip on D1, 28 days a cycle.
  Other Names: PDR001

SUMMARY:
This study examines the safety and efficacy of ribociclib (CDK 4/6 inhibitors) and spartalizumab (anti-PD1) in patients with recurrent and/or metastatic head and neck squamous cell carcinoma (R/M HNSCC).

DETAILED DESCRIPTION:
The study is a phase I study testing ribociclib (with dose titration plan) and spartalizumab (fixed dose) for R/M HNSCC. The primary endpoints are safety and objective response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of oral cavity, oropharynx, hypopharynx, or larynx.
2. The recurrent disease is not suitable for curative surgery or definitive chemoradiation, and/or metastatic diseases which are not amenable to surgery and/or curative radiotherapy.
3. Measurable disease according to RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
4. Age: older than 20 years-old, and younger than 70 years-old
5. ECOG performance status: ≤ 1
6. Adequate organ function,
7. Recovered from any previous therapy related toxicity to ≤Grade 1 at study entry (except for stable sensory neuropathy ≤Grade 2 and alopecia)
8. Patient must have the following laboratory values within local normal range or corrected to within local normal range with supplements before the first dose of study medication:

   * Sodium
   * Potassium
   * Magnesium
   * Total Calcium (corrected for serum albumin)
   * Phosphorus
9. Standard 12-lead ECG values defined as the mean of the triplicate ECGs and assessed by the local laboratory

   * QTcF interval at screening < 450 msec (using Fridericia's correction)
   * Mean resting heart rate 50-100 bpm (determined from the ECG)
10. Agree to take biopsy before and during the treatment
11. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
12. Female subject of childbearing potential should have a negative urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) OR
    2. A WOCBP who agrees to have the contraceptive during the treatment period and for at least 120 days after the last dose of study treatment
14. A male participant must agree to use a contraception of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

1. Nasopharyngeal carcinoma or nasal cavity malignancies other than HNSCC
2. For patients with oropharyngeal cancer, positive p16 immunohistochemical (IHC) stain is excluded.

   The positivity of p16 IHC is defined as p16 IHC expression ≥ 70
3. Concurrent malignancies other than HNSCC
4. Can not take a complete tablet orally.
5. Hypercalcemia [corrected serum calcium > upper limits of normal (ULN)] in recent 42 days.
6. Prior exposure to anti-PD-1, anti-PD-L1, anti-CTLA-4, or other immune checkpoint inhibitors
7. Prior exposure to ribociclib, palbociclib, or abemaciclib.
8. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as detectable HCV RNA) infection.
9. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
10. Has an active infection requiring systemic therapy 14 days before signing informed consent.
11. Has received prior radiotherapy within 4 weeks of signing informed consent.
12. Major surgery within 4 weeks before signing informed consent.
13. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of ≥ 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to signing informed consent.
14. Has known history of pneumonitis requiring steroids, or any evidence of active, non-infectious pneumonitis, or other known interstitial lung disease
15. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
16. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Topical or inhaled steroids is not considered as systemic treatment.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug
20. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
21. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
22. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhoea, malabsorption)
23. Known brain metastases or leptomeningeal carcinomatosis
24. History of severe hypersensitivity reactions to other monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 28 days
  CTCAE 5.0
Objective response rate | 8 weeks
  RECIST 1.1

SECONDARY OUTCOMES:
Progression free survival | 24 months
  from study entry to disease progression or death
Overall survival | 24 months
  from study entry to death
Duration of response | 24 months
  from response to disease progression
Objective response rate (iRECIST) | 8 weeks
  iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Fong Kao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No